CLINICAL TRIAL: NCT01371539
Title: Clinical Comparison of Two Multifocal Contact Lenses Made of Silicone Hydrogel Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-319-C-021
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-06

CONDITIONS: Myopia; Presbyopia
Keywords: Myopia; Presbyopia
MeSH Terms: conditions — Myopia; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon B / Comfilcon A (Other): Lotrafilcon B contact lenses worn first, with comfilcon A contact lenses worn second. Both products worn bilaterally on a daily wear basis for one week each.
  Interventions: Device: Lotrafilcon B contact lens; Device: Comfilcon A contact lens
- Comfilcon A / Lotrafilcon B (Other): Comfilcon A contact lenses worn first, with lotrafilcon B contact lenses worn second. Both products worn bilaterally on a daily wear basis for one week each.
  Interventions: Device: Lotrafilcon B contact lens; Device: Comfilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon B contact lens — Commercially marketed, silicone hydrogel, multifocal contact lens for daily wear use.
  Other Names: AIR OPTIX AQUA MULTIFOCAL
Device: Comfilcon A contact lens — Commercially marketed (France), silicone hydrogel, multifocal contact lens for daily wear use.
  Other Names: Biofinity Multifocal

SUMMARY:
The purpose of this study was to compare visual performance measures between two multifocal contact lenses on presbyopic wearers.

ELIGIBILITY:
Inclusion Criteria:

* At least 35 years of age.
* Spectacle add of +0.50 to +2.50 diopters (inclusive).
* Currently wearing soft contact lenses at least 5 days per week and at least 8 hours per day.
* Able to be fit in both eyes with soft multifocal lenses in available powers.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within 12 weeks of enrollment in trial.
* Currently enrolled in any clinical trial.
* Astigmatism of 1.00 diopter or more.
* Currently wearing excluded brands of multifocal lenses, as specified by protocol.
* Other protocol-defined exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Cummings, O.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from 12 US private practices.
Pre-assignment Details: Five participants were enrolled, but not dispensed, due to failing inclusion/exclusion criteria (4) and unacceptable subjective vision (1). Baseline characteristics are presented on all enrolled and dispensed participants: 104.
Period: Period One: One Week
Arm/Group | Lotrafilcon B / Comfilcon A | Comfilcon A / Lotrafilcon B
Started | 53 | 51
Completed | 53 | 50
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Period Two: One Week
Arm/Group | Lotrafilcon B / Comfilcon A | Comfilcon A / Lotrafilcon B
Started | 53 | 50
Completed | 53 | 47
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Unacceptable Objective Visual Acuity | 0 | 1
Not completed — Time/job conflict | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: All enrolled and dispensed participants
Arm/Group | Overall
Number analyzed (Participants) | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 49.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 104

OUTCOME MEASURES:

1. Primary Outcome: Corrected Distance Binocular Visual Measurement in Normal Illumination Reported as Binocular Distance Visual Acuity
Description: The participant read a Snellen chart at a 20-foot equivalent distance with both eyes together while wearing study lenses. The Snellen acuity was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equated to a logMAR acuity of 0.0 and was considered normal distance eyesight. A positive logMAR value indicated poorer vision, and a negative value denoted better visual acuity.
Time Frame: 1 week
Population: The Efficacy Evaluable Set (EES) contained all enrolled and dispensed subjects with no major protocol deviations as determined by masked review that also completed a minimum of 4 days of lens wear with either study product and attended an assessing follow-up visit.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Lotrafilcon B: Lotrafilcon B contact lenses worn bilaterally on a daily wear basis for one week.
- Comfilcon A: Comfilcon A contact lenses worn bilaterally on a daily wear basis for one week.
Arm/Group | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 98 | 101
logMAR | -0.00 (0.07) | 0.00 (0.06)

2. Primary Outcome: Corrected Near Binocular Visual Measurement in Normal Illumination Reported as Binocular Near Visual Acuity
Description: The participant read a Snellen chart at 40 centimeters with both eyes together while wearing study lenses. The Snellen acuity was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equated to a logMAR acuity of 0.0 and was considered normal near eyesight. A positive logMAR value indicated poorer vision, and a negative value denoted better visual acuity.
Time Frame: 1 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 98 | 102
logMAR | 0.12 (0.10) | 0.10 (0.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 24-JUN-2011 to 16-AUG-2011.
Description: The safety population included all enrolled and dispensed participants. One participant was dispensed the control product only in this cross-over study.
Arm/Group | Lotrafilcon B | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/104
Other Adverse Events (participants affected / at risk) | 0/103 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.